CLINICAL TRIAL: NCT02884921
Title: Preemptive Analgesia Using Intravenous Paracetamol in Dental Sitting
Brief Title: Preemptive Analgesia Using Intravenous Paracetamol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, MD, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-008
Record Dates: First submitted 2016-08-21; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Postoperative pain; Dental treatment; Paracetamol
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preemptive Paracetamol (Active Comparator): Preemptive Paracetamol
  Interventions: Drug: Paracetamol
- Post surgery Paracetamol (Active Comparator): Post surgery Paracetamol
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Paracetamol
  Arms: Preemptive Paracetamol
Drug: Paracetamol — Paracetamol
  Arms: Post surgery Paracetamol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Dental treatment for children should be done in a calm atmosphere and without pain. Oral Propacetamol has been shown to be effective in a variety of postsurgical pain models.

There are no studies on paracetamol preemptive analgesia effect on the pediatric population in the dental setting which compare analgesic effect when administered before Vs after the dental treatment.

The investigators hypothesis is that preoperative intravenous paracetamol are helpful in the prevention of postoperative pain in children undergoing dental treatment.

DETAILED DESCRIPTION:
Dental treatment for children should be done in a calm atmosphere and without pain in purpose to achieve a positive feelings and response towards dental treatment.Postoperative pain is the main issue which may cause a negative attitude of the child to dental treatment in future appointment. One of the affective options to deal with this pain is to give analgesic drug before the initiative of treatment which should continue its effect during and may also after treatment which is known as "preemptive analgesia. Oral Propacetamol has been shown to be effective in a variety of postsurgical pain models. In double blind clinical trials single or multiple dose of intravenous paracetamol, generally provided significantly better analgesic effect than placebo treatment in adults' patients who had undergone dental, orthopedic or gynecological surgery. There is considerable evidence that the analgesic effect of paracetamol is central and is due to activation of descending serotonergic pathways, but its primary site of action may still be inhibition of prostaglandin synthesis by its selective inhibition of Cox-2 isoenzyme.

At the best of the investigators knowledge, there are no studies on paracetamol preemptive analgesia effect on the pediatric population in the dental setting which compare analgesic effect when administered before Vs after the dental treatment.

The investigators hypothesis is that preoperative intravenous paracetamol are helpful in the prevention or modification of postoperative pain in children undergoing dental treatment.

The primary outcome of this study is to investigate the post dental treatment analgesic effect of intravenous paracetamol in children when administered before compared to after dental treatment.

ELIGIBILITY:
Inclusion criteria:

* All children who require a wide treatment of caries
* Children of high score of anxious or who is stressfully

Exclusion criteria:

* Contraindication for paracetamol
* Renal or hepatic insufficiency
* Patient have history of allergy for paracetamol
* Anemia of Hgb less than 10 gr/DL

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain measure in numerical scale | 1-24 hours
  Post operative Pain measure in numerical scale from 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: mira koch, Study Chair — Ethicla Committee Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes